CLINICAL TRIAL: NCT03966053
Title: Phase I/II, Open Label Study to Determine Safety of Trifluoperazine (TFP) in Adults With Red Blood Cell Transfusion-Dependent Diamond Blackfan Anemia
Brief Title: The Use of Trifluoperazine in Transfusion Dependent DBA
Acronym: DBA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Supporter terminated study due to slow subject accrual secondary to COVID pandemic limiting travel to research site.
Sponsor: Adrianna Vlachos, MD (Other)
Responsible Party: Sponsor-Investigator, Adrianna Vlachos, MD, Head, Bone Marrow Failure Program, Feinstein Institute for Medical Research
Organization: Northwell Health (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-0748
Record Dates: First submitted 2019-05-23; First posted 2019-05-29 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Diamond Blackfan Anemia; Pure Red Cell Aplasia
Keywords: Diamond Blackfan Anemia
MeSH Terms: conditions — Anemia, Diamond-Blackfan; Red-Cell Aplasia, Pure | interventions — Trifluoperazine

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Cohort A: Three subjects will receive Trifluoperazine (TFP) 1 mg PO daily.
  * If there is no non-neurologic toxicity Grade 3 at the end of the 21 days, Cohort B will start.
  * If 1/3 subjects in Cohort A demonstrates toxicity Grade 3, an additional 3 subjects will be enrolled in Cohort A.
  * If 2 or more of the 6 subjects in Cohort A demonstrate toxicity Grade 3, the trial will be stopped; no MTD will be declared.
  * If less than 2 of the 6 subjects in Cohort A demonstrate toxicity Grade 3 within 21 days of starting therapy, Cohort B will start.
  Interventions: Drug: Trifluoperazine
- Cohort B (Experimental): Cohort B: Three subjects will receive TFP 2 mg PO daily.
  * If there is no non-neurologic toxicity Grade 3 at the end of the 21 days, Cohort C will start.
  * If 1/3 subjects in Cohort B demonstrates toxicity Grade 3, an additional 3 subjects will be enrolled in Cohort B:
  * If 2 or more of the 6 subjects in Cohort B demonstrate toxicity Grade 3, the study will be stopped, and 1 mg/day will be declared the MTD.
  * If < 2 of the 6 subjects in Cohort B demonstrate toxicity Grade 3 within 21 days of starting therapy, Cohort C will start.
  Interventions: Drug: Trifluoperazine
- Cohort C (Experimental): Cohort C: Three subjects will receive TFP 5 mg PO daily.
  * If there is no non-neurologic toxicity ≥ Grade 3 at the end of the 21 days, Cohort D will start.
  * If 1/3 subjects in Cohort C demonstrates toxicity Grade 3, an additional 3 subjects will be enrolled in Cohort C:
  * If 2 or more of the 6 subjects in Cohort C demonstrate toxicity Grade 3, the study will be stopped, and 2 mg/day will be declared the MTD.
  * If < 2 of the 6 subjects in Cohort C demonstrate toxicity Grade 3 within 21 days of starting therapy, cohort D will start.
  Interventions: Drug: Trifluoperazine
- Cohort D (Experimental): Cohort D: Three subjects will receive TFP 10 mg PO daily.
  * If 0/3 subjects in Cohort D demonstrates toxicity Grade 3, the study will be stopped, and 10 mg/day will be declared the MTD.
  * If 1/3 subjects in Cohort D demonstrates toxicity Grade 3, an additional 3 subjects will be enrolled in Cohort D.
  * If 2 or more of the 6 subjects in Cohort D demonstrate toxicity Grade 3, the study will be stopped, and 5 mg/day will be declared the MTD.
  * If <2 of the 6 subjects in Cohort D demonstrate toxicity > Grade 3 within 21 days of starting therapy, 10mg/day will be declared the MTD.
  Interventions: Drug: Trifluoperazine

INTERVENTIONS:
Drug: Trifluoperazine — Trifluoperazine (TFP)1mg, 2mg, 5mg, or 10mg will be given once daily by mouth for 21 days
  Other Names: TFP

SUMMARY:
Diamond Blackfan anemia (DBA) is a rare inherited pure red cell aplasia. The two main non-stem cell transplant therapeutic options are corticosteroids and red blood cell (RBC) transfusions. About 80% of DBA patients initially respond to corticosteroids, however, half of the patients cannot continue due to side effects or loss of response. These patients are then typically dependent on RBC transfusions throughout life. Each of these treatments is fraught with many side effects and significant morbidity and mortality are potential consequences of hematopoietic stem cell transplantation (SCT). The majority of individuals with DBA have mutations in genes encoding structural proteins of the small or large ribosomal subunit leading to deficiency of the particular ribosomal protein (RP). Using the RP deficient zebrafish embryo model, high throughput drug screens have demonstrated a strong hematologic response to several calmodulin inhibitors. One of these chemicals is trifluoperazine (TFP). TFP treatment of a mouse model of DBA also increased the red blood cell count and the hemoglobin (Hb) levels in the mice. TFP is a FDA-approved typical antipsychotic agent that has been available since 1958 with a well-known safety profile. In the United States, TFP is approved for the short-term treatment of generalized non-psychotic anxiety; treatment or prevention of nausea and vomiting of various causes; and, management of psychotic disorders.

This study aims to determine the safety/tolerability of TFP in adult subjects with DBA. TFP's expected dose-limiting toxicity is primarily neurologic (extrapyramidal) when used long-term at typical anti-psychotic doses (range 10-50 mg daily). Non-neurologic adverse effects in subjects with DBA have not been investigated. We will perform a dose escalation study to define the safety and tolerability of lower doses of this agent in subjects with DBA. To mitigate the potential risks of administering TFP to this new population, we will (1) start dosing at dose levels well below those prescribed for psychosis, (2) dose escalate to a maximum of 10 mg daily (the lowest dose typically prescribed for psychosis), and (3) perform weekly safety monitoring. Given the positive signal in DBA animal models and the 60-year clinical experience with higher doses of TFP, this drug warrants a trial in humans to assess tolerability in DBA.

DETAILED DESCRIPTION:
This is a dose escalation safety/tolerability study to evaluate the presence of TFP-related adverse events in DBA subjects, and to determine the maximum tolerated dose (MTD) of TFP in DBA.

If tolerated, this trial will support either a proof of concept trial of low-dose TFP in DBA, or the advancement of a chemically modified TFP-like drug (to alleviate the neurologic toxicity) for the treatment of DBA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age: 18 years and <65 years of age.
* Weight: ≥45 kilograms.
* DBA diagnosed according to the DBA criteria (Vlachos, 2008)
* RBC transfusion-dependence (defined as 2 units packed RBCs per 28 days averaged over 84 days [12 weeks] prior to study entry)
* Calculated creatinine clearance > 30 mL/min
* Karnofsky performance status scale score ≥ 70
* Female subjects of childbearing potential must have a negative serum pregnancy test and use highly effective methods of birth control during the study
* Male subjects must agree to use a latex condom during any sexual contact with females of childbearing potential while participating in the study
* Agreement to adhere to the study visit schedule, understand and comply with all protocol requirements.

Exclusion Criteria:

* Liver: aspartate aminotransferase (AST) > 5 x the upper limit of normal (ULN), alanine aminotransferase (ALT) >5 x ULN, or bilirubin > 5 x ULN
* Heart disease (New York Heart Association classification of ≥ 3)
* History of angina
* Uncontrolled hypertension
* Subjects currently responsive to corticosteroids for treatment of DBA.
* Treatment with another investigational drug or device <56 days pre-study entry.
* Pregnant or lactating females
* Any history of severe allergic reaction requiring the use of epinephrine
* Known hypersensitivity to the study drug or other phenothiazines
* History or presence of extrapyramidal signs
* History of cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrianna Vlachos, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Boston Children's hospital, Boston, Massachusetts
  - The Feinstein Institute for Medical Research, Manhasset, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Cohort A: Three subjects will receive Trifluoperazine (TFP) 1 mg PO daily.
  * If there is no non-neurologic toxicity Grade 3 at the end of the 21 days, Cohort B will start.
  * If 1/3 subjects in Cohort A demonstrates toxicity Grade 3, an additional 3 subjects will be enrolled in Cohort A.
  * If 2 or more of the 6 subjects in Cohort A demonstrate toxicity Grade 3, the trial will be stopped; no MTD will be declared.
  * If less than 2 of the 6 subjects in Cohort A demonstrate toxicity Grade 3 within 21 days of starting therapy, Cohort B will start.
  Trifluoperazine: Trifluoperazine (TFP)1mg, 2mg, 5mg, or 10mg will be given once daily by mouth for 21 days
Period: Overall Study
Arm/Group | Cohort A
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by subject prior to starting study drug. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cohort A
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by the Simpson-Angus Scale and CTCAE v4.0
Description: Each subject will undergo weekly safety assessment using the Simpson-Angus Extrapyramidal Side Effects Scale to determine the safety of TFP in this new population of patients. The subjects will also undergo weekly bloodwork to evaluate for any liver or kidney abnormalities as well as a complete blood count and reticulocyte count. All dosed subjects will be followed for an additional 1 week after discontinuing study drug (post-study safety follow-up). There will be no more than 6 subjects enrolled at any particular time.
  Treatment will be discontinued for any subject if their Hb is > 12 gm/dL , and not associated with RBC transfusions.
Time Frame: The subjects will be evaluated weekly for 4 weeks after the start of the 21-day course, 3 weeks while on the study drug and one week after completion.
Population: One subject received study drug. The other subject did not receive study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Cohort A
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Protocol closed early due to slow accrual secondary to COVID travel restrictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT03966053/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT03966053/ICF_000.pdf